CLINICAL TRIAL: NCT00550823
Title: The Use of Cardiac Computarized Tomography in Infective Endocarditis
Brief Title: Cardiac Computarized Tomography in Infective Endocarditis
Acronym: cardiac CT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 362-07
Record Dates: First submitted 2007-10-27; First posted 2007-10-30 (Estimated); Last update posted 2007-10-30 (Estimated); Status verified 2007-10

CONDITIONS: Infective Endocarditis
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A,1 (Experimental)
  Interventions: Device: Cardiac CT 0BRILLIANT 64

INTERVENTIONS:
Device: Cardiac CT 0BRILLIANT 64 — Cardiac CT

SUMMARY:
The diagnosis of infective endocarditis is based on the results of blood culture and findings on transeosophageal echocardiography. Cardiac computarized tomography is a new modality, mainly used for the imaging of coronary arteries. Its use in the diagnosis of infective endocarditis is not well known.The purpose of this study is to establish the use of cardiac CT in infective endocarditis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with infective endocarditis

Exclusion Criteria:

* Allergy to contrast agent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-11; Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
The diagnostic capacity of cardiac CT in comparison with TEE in the diagnosis of infective endocarditis | 1 year

SECONDARY OUTCOMES:
Assessment of cardiac function in patients with infective endocarditis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ori Elkayam, M.D, Principal Investigator — Tel Aviv Medical Center